CLINICAL TRIAL: NCT05535829
Title: Molecular Markers in Predicting Response to Treatment in FH-deficient RCC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Tongji Hospital (Other); Changzhou No.2 People's Hospital (Other); Ruijin Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai 10th People's Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Shanghai Zhongshan Hospital (Other); Jiangxi Provincial People's Hopital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Zhejiang Provincial People's Hospital (Other); Peking University First Hospital (Other); Zhejiang University (Other); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: RENJIFHRCC
Record Dates: First submitted 2022-08-15; First posted 2022-09-10 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: FH-Deficient RCC; Systemic Treatments; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with FH-deficient RCC: Laboratory analysis of samples
  Interventions: Other: Laboratory analysis of samples

INTERVENTIONS:
Other: Laboratory analysis of samples — Laboratory analysis of samples

SUMMARY:
Fumarate hydratase-deficient renal cell carcinoma (FH-deficient RCC) is a rare subtype of RCC characterized by germline/somatic mutation of the fumarate hydratase (FH) gene, and is an extremely aggressive tumor, with a propensity to disseminate early even in the setting of a small primary tumor. This project is a real-world exploratory study aiming to explore potential molecular markers detectable at baseline that can enable the prediction of clinical efficacy of systemic treatments in advanced FH-deficient RCC.

This project is a real-world exploratory study aiming to explore potential molecular markers detectable at baseline that can enable the prediction of clinical efficacy of immunotherapy combined with target therapy in advanced FH-deficient RCC.

This study aims to include a total of 100 patients initially diagnosed with advanced FH-deficient RCC. Paired tissue and blood samples collected from all patients before or/ and after the start of immunotherapy-based treatment (at diagnosis or/ and their change with treatment) will be analyzed.

The patient samples will be submitted for molecular analysis, including next-generation sequencing (NGS)-based gene expression profiling (GEP), RNA-sequencing, multiplex immunofluorescence staining and inflammation-related T-cell receptor (TCR) repertoire profiling, ect. The molecular assay results will include but will not be limited to tumor mutation burden (TMB), microsatellite instability (MSI) status, DNA damage repair (DDR)-related gene mutation status, and programmed death-ligand 1 (PD-L1) expression level. Patients will be followed-up for treatment responses until radiological confirmation of disease progression to immunotherapy-based treatment. The molecular assay results will then be analyzed with clinical data including objective responses and progression-free survival outcomes, among others, to identify molecular markers at baseline that are associated with clinical efficacy of immunotherapy-based treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. histopathological evidence of FH-deficient RCC, which was confirmed by Sanger or next-generation sequencing after initial screening by IHC.
3. included patients must be diagnosed with metastatic renal cell carcinoma or have a TNM stage IV (according to 2009 TNM Classification);
4. new FH-deficient RCC patients who has scheduled to start 1st cycle of systemic treatment;
5. ECOG score ≤2;
6. life expectancy ≥ 3 months;
7. sign informed consent, and be able to follow the visit and related procedures stipulated in the program;
8. agree to collect tumor tissue, blood and other specimens required by this study and apply them to relevant studies;

Exclusion Criteria:

1. patients with other malignant tumors with different primary sites or histology from the tumor evaluated in this study within 2 years of personal history.
2. major surgery or severe trauma within 4 weeks before enrollment;
3. known or suspected active autoimmune diseases (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. Patients with type 1 diabetes with good insulin control can also be enrolled.
4. known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
5. allergic to any component of monoclonal antibody;
6. suffering from other uncontrolled serious diseases, including but not limited to: A) severe infection in the active phase or clinically poorly controlled; B) HIV infection (HIV antibody positive); C) acute or chronic active hepatitis b (HBsAg positive and HBV DNA>1*103/ml) or acute or chronic active hepatitis c (HCV antibody positive and HCV RNA>15IU/ml); D) active tuberculosis, etc.;
7. class iii-iv congestive heart failure (New York heart association classification), poorly controlled and clinically significant arrhythmia;
8. uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg);
9. pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced FH-deficient RCC who have given prior consent for their samples and data to be used, and who have received immunotherapy-based treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Systemic treatment OS | Through study completion, an average of 3 year
  Systemic treatment OS was defined as the time from the start of systemic treatment to death from any cause, and patients without a recorded death were right censored to the date of last clinical visit or clinical record.

SECONDARY OUTCOMES:
First-line PFS | Through study completion, an average of 3 year
  First-line progression free survival (PFS) was defined as the time from the start of first-line systemic treatment to the time of radiographic progression, or death from any cause, whichever occurred first.
ORR | Through study completion, an average of 3 year
  Objective response rate (ORR) was defined as complete response (CR)+ partial response (PR)
DCR | Through study completion, an average of 3 year
  disease control rate (DCR) was defined as partial response (PR)+complete response (CR)+stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No